CLINICAL TRIAL: NCT05223010
Title: Evaluation of Preoperative Melatonin on Emergence Agitation After Herniorrhaphy Surgeries in Pediatrics
Brief Title: Melatonin for Pediatric Emergence Agitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1/2022ANET3-A
Record Dates: First submitted 2022-01-07; First posted 2022-02-03 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Emergence Agitation
Keywords: melatonin; emergence agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Melatonin; Solutions; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Active Comparator): 39 participant will receive melatonin 0.05 mg/kg
  Interventions: Drug: Melatonin 5 MG/15 ML Oral Solution 0.05 mg/kg; Drug: Sevoflurane
- 2 (Active Comparator): 39 participant will receive melatonin 0.2 mg/kg
  Interventions: Drug: Melatonin 5 MG/15 ML Oral Solution 0.2mg/kg; Drug: Sevoflurane
- 3 (Active Comparator): 39 participant will receive melatonin 0.4 mg/kg
  Interventions: Drug: Melatonin 5 MG/15 ML Oral Solution 0.4mg/kg; Drug: Sevoflurane

INTERVENTIONS:
Drug: Melatonin 5 MG/15 ML Oral Solution 0.05 mg/kg — will be administered 1 hour before arrival to operating room
  Arms: 1
Drug: Melatonin 5 MG/15 ML Oral Solution 0.2mg/kg — will be administered 1 hour before arrival to operating room
  Arms: 2
Drug: Melatonin 5 MG/15 ML Oral Solution 0.4mg/kg — will be administered 1 hour before arrival to operating room
  Arms: 3
Drug: Sevoflurane — for anaesthesia induction 3-8 MAC

SUMMARY:
efficacy of melatonin premedication on emergence agitation in children undergoing herniorrhaphy surgeries

DETAILED DESCRIPTION:
Before administration of the oral premedication, each patient's baseline heart rate, mean systemic arterial pressure, pulse oximetry, and sedation score (yale preoperative score) will be recorded All the anesthetic and surgical techniques will be standardized. On arrival at the operating room, continuous electrocardiogram, non-invasive blood pressure and pulse oximetry monitors will be applied. Baseline readings of all the parameters will be recorded.

Sevoflurane 3-8 MAC will be used for induction of anaesthesia. While intravenous line is inserted, atropine 0.01 mg/kg, atracurium 0.0.05 mg/kg is given. Anaesthesia maintainance done by 1.5-2 MAC sevoflurane. At the end of operation discontinuation of inhalational anesthesia will be done and muscle relaxant will be reversed by neostigmine 0.05 mg/kg and atropine 0.02 mg/kg. Then children were transferred to recovery till complete recovery Parameters assessed are induction time (IT) time from the start of sevoflurane inhalation to the start of endtracheal tube insertion, duration of anesthesia (DA) time from the start of sevoflurane inhalation to discontinuation of sevoflurane inhalation, time up to spontaneous eye opening (time from removal of endotracheal tube till spontaneous eye opening), duration of stay in recovery and any side effects

ELIGIBILITY:
Inclusion Criteria:

* ASA I
* scheduled for unilateral inguinal herniorrhaphy
* parents conscent

Exclusion Criteria:

* allergy to this study drug
* Patients with a history of cardiovascular, psychiatric, neurological, endocrine, chest disease, and/or severe renal or hepatic dysfunction

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — inguinal hernia is common in males
Enrollment: 117 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
emergence behaviour | 5 min, 15 min and 30 min after arrival to recovery
  change from baseline on a 5 point scale

SECONDARY OUTCOMES:
yale preoperative anxiety scale | before administration of oral premedication and before anaesthesia induction
  3 domain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University Hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No